CLINICAL TRIAL: NCT00963976
Title: Intracerebral Hemorrhage Acutely Decreasing Arterial Pressure Trial
Acronym: ICH ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Principal Investigator, Ken Butcher, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICHADAPT513000128
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Intracerebral Hemorrhage
Keywords: Stroke; Hypertension; Cerebral Blood Flow; CT Perfusion
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hypertension | interventions — Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Target systolic BP < 150 mmHg (Experimental): Systolic blood pressure will be reduced to <150 mmHg within 1 hour of randomization.
  Interventions: Drug: labetalol/hydralazine/enalapril
- Target systolic BP < 180 mmHg (Active Comparator): Systolic blood pressure will be reduced, to <180 mmHg within 1 hour of randomization.
  Interventions: Drug: labetalol/hydralazine/enalapril

INTERVENTIONS:
Drug: labetalol/hydralazine/enalapril — Blood pressure will be treated with intravenous labetalol (10 mg starting dose)/hydralazine (5 mg starting dose)/enalapril (1.25 mg starting dose).

SUMMARY:
Rationale: Management of blood pressure (BP) in the acute phase of intracerebral hemorrhage (ICH) remains controversial. Although it has been established that there is a transient moderate reduction of perihematoma cerebral blood flow (CBF) in acute ICH, the effect of BP treatment is unknown. The potential for exacerbation of CBF has precluded routine aggressive BP reduction.

Aim and Hypothesis: The primary study aim is to demonstrate the feasibility and safety of acute BP reduction to < 150 mmHg systolic using a standardized protocol in ICH patients. It is hypothesized that CTP will not demonstrate evidence of perihematoma ischemia following acute BP reduction.

Design: ICH ADAPT is a randomized blinded endpoint trial. Acutely hypertensive ICH patients are randomized to a target systolic BP of < 150 mmHg or < 180 mmHg. Patients are treated with intravenous (IV) labetalol/hydralazine/enalapril.

Study Outcomes: The primary outcome is cerebral blood flow in the perihematoma region, measured with CT perfusion, 2 hours after randomization. Secondary outcomes include the difference in BP at 1 and 2 hours post-randomization in the two treatment groups and hematoma expansion rates at 24 hours.

Discussion: ICH ADAPT is the only randomized trial designed specifically to identify any hemodynamic changes in the perihematoma region secondary to aggressive BP management. The results of this trial will facilitate ongoing and future studies aimed at determining the efficacy of rapid BP reduction in acute ICH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute primary ICH demonstrated with CT scan
* Onset ≤ 24 h prior to randomization

Exclusion Criteria:

* Contraindication to BP reduction i.e., severe arterial stenosis or high-grade stenotic valvular heart disease
* Indication for urgent BP reduction i.e., hypertensive encephalopathy, or aortic dissection
* Definite evidence that the ICH is secondary to underlying cerebral or vascular pathology, i.e., AVM, aneurysm, tumour, trauma, vasculitis, or hemorrhagic transformation of an ischemic infarct
* Previous ischemic stroke within 30 days of current event NB: Prior ICH is not an exclusion criterion
* Planned surgical resection of hematoma NB: Extraventricular Drain placement is not an exclusion criterion
* Contraindication to CT perfusion imaging (i.e. contrast allergy, metformin use or Creatinine >160 μmol/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is cerebral blood flow in the perihematoma region, measured with CT perfusion, 2 hours after randomization. | 2 hours post randomization

SECONDARY OUTCOMES:
Hematoma expansion rates at 24 hours. | 24 hours post randomization

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - University of Ottawa, Ottawa, Ontario

REFERENCES:
- [Derived] Klahr AC, Kosior JC, Dowlatshahi D, Buck BH, Beaulieu C, Gioia LC, Kalashyan H, Wilman AH, Jeerakathil T, Emery DJ, Shuaib A, Butcher KS. Lower Blood Pressure Is Not Associated With Decreased Arterial Spin Labeling Estimates of Perfusion in Intracerebral Hemorrhage. J Am Heart Assoc. 2019 Jun 4;8(11):e010904. doi: 10.1161/JAHA.118.010904. PMID 31131671
- [Derived] McCourt R, Gould B, Kate M, Asdaghi N, Kosior JC, Coutts S, Hill MD, Demchuk A, Jeerakathil T, Emery D, Butcher KS. Blood-brain barrier compromise does not predict perihematoma edema growth in intracerebral hemorrhage. Stroke. 2015 Apr;46(4):954-60. doi: 10.1161/STROKEAHA.114.007544. Epub 2015 Feb 19. PMID 25700288
- [Derived] Gould B, McCourt R, Gioia LC, Kate M, Hill MD, Asdaghi N, Dowlatshahi D, Jeerakathil T, Coutts SB, Demchuk AM, Emery D, Shuaib A, Butcher K; ICH ADAPT Investigators. Acute blood pressure reduction in patients with intracerebral hemorrhage does not result in borderzone region hypoperfusion. Stroke. 2014 Oct;45(10):2894-9. doi: 10.1161/STROKEAHA.114.005614. Epub 2014 Aug 21. PMID 25147326
- [Derived] McCourt R, Gould B, Gioia L, Kate M, Coutts SB, Dowlatshahi D, Asdaghi N, Jeerakathil T, Hill MD, Demchuk AM, Buck B, Emery D, Butcher K; ICH ADAPT Investigators. Cerebral perfusion and blood pressure do not affect perihematoma edema growth in acute intracerebral hemorrhage. Stroke. 2014 May;45(5):1292-8. doi: 10.1161/STROKEAHA.113.003194. Epub 2014 Apr 1. PMID 24692481
- [Derived] Butcher KS, Jeerakathil T, Hill M, Demchuk AM, Dowlatshahi D, Coutts SB, Gould B, McCourt R, Asdaghi N, Findlay JM, Emery D, Shuaib A; ICH ADAPT Investigators. The Intracerebral Hemorrhage Acutely Decreasing Arterial Pressure Trial. Stroke. 2013 Mar;44(3):620-6. doi: 10.1161/STROKEAHA.111.000188. Epub 2013 Feb 7. PMID 23391776
- [Derived] Butcher K, Jeerakathil T, Emery D, Dowlatshahi D, Hill MD, Sharma M, Buck B, Findlay M, Lee TY, Demchuk AM. The Intracerebral Haemorrhage Acutely Decreasing Arterial Pressure Trial: ICH ADAPT. Int J Stroke. 2010 Jun;5(3):227-33. doi: 10.1111/j.1747-4949.2010.00431.x. PMID 20536619